CLINICAL TRIAL: NCT02649816
Title: A Retrospective Cohort Study on Clinical Success of Resin Sealants
Brief Title: Effectiveness of Resin Sealants: Retrospective Cohort Study
Status: Completed | Type: Observational
Sponsor: Fernanda Miori Pascon (Other)
Responsible Party: Sponsor-Investigator, Fernanda Miori Pascon, Teacher, University of Campinas, Brazil
Organization: University of Campinas, Brazil (Other)
Other Study IDs: 2
Record Dates: First submitted 2015-12-23; First posted 2016-01-07 (Estimated); Last update posted 2016-01-07 (Estimated); Status verified 2016-01

CONDITIONS: Dental Caries
Keywords: Pit and fissure sealants; Dental Caries; Prevention; Dental undergraduate students; patient's caries risk
MeSH Terms: conditions — Dental Caries; Van der Woude syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This retrospective cohort study assessed sealant clinical success applied to pit and fissure by dental undergraduate students at Piracicaba Dental School - Brazil.

DETAILED DESCRIPTION:
A population presenting 1st/2nd permanent molars with sealed occlusal surfaces were considered. Dental records were reviewed for: patient's caries risk (High/Low); operator experience (scores 1 to 4, beginners to seniors); number of follow-up visits; isolation procedure; sealant/tooth type; and age at placement. Posteriorly, the patients were called to dental evaluation and the sealed teeth were classified regarding the sealant presence, partial presence or absence, with or without caries, or sealant replacement to a restorative material in Satisfactory or Unsatisfactory, considering the caries presence/absence. Successful outcome was considered in the caries absence.

ELIGIBILITY:
Inclusion Criteria:

* A population presenting first and second permanent molars with sealed occlusal surfaces by dental undergraduate students at Piracicaba Dental School Brazil.

Exclusion Criteria:

* First and second permanent molars with sealed occlusal surfaces by dentistry.

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Patients treated at Piracicaba Dental School - Brazil
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2011-03; Primary Completion 2012-03 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Probability (%) of the caries development in the treated teeth assessed by Kaplan-Meier survival analysis (Bioestat 5.3). | 1 year
  Outcome mensuration by clinical examination (caries prevention and retention sealant) and bitewing radiograph.

CONTACTS AND LOCATIONS:
Overall Officials: Juliana Camargo, Principal Investigator — Piracicaba Dental School - University of Campinas; Kelly Moreira, Principal Investigator — Piracicaba Dental School - University of Campinas

IPD SHARING:
Plan to Share IPD: No